CLINICAL TRIAL: NCT05935345
Title: Addressing Nonsuicidal Self-injury in Schools
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Östergötland (Other)
Responsible Party: Principal Investigator, Maria Zetterqvist, Principal investigator, Region Östergötland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021-01699
Record Dates: First submitted 2023-04-30; First posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Nonsuicidal Self-injury; Suicidal Ideation; Stigmatization; Help-Seeking Behavior; Perceived Social Support; Mental Well-being
Keywords: Prevention; Whole-school approach; Nonsuicidal self-injury; Suicidality; Stigma; Help-seeking; Mental health
MeSH Terms: conditions — Self-Injurious Behavior; Suicidal Ideation; Stereotyping; Help-Seeking Behavior; Psychological Well-Being; Social Stigma | interventions — Schools

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Addressing NSSI in schools (Experimental): During the four months of active experimental condition, adolescents receive five sessions of the youth aware of mental health program in the class room, and one additional session on NSSI. Parents and school staff receive an online psychoeducation on NSSI. School health care personnel receive a 2-day workshop on NSSI and suicidality.
  Interventions: Behavioral: Addressing NSSI in schools
- Control condition (Other): Participating adolescents, parents, teachers and school health care personnel receive no intervention during four months
  Interventions: Other: Control condition

INTERVENTIONS:
Behavioral: Addressing NSSI in schools — During the four months of active experimental condition, adolescents receive five sessions of the youth aware of mental health program in the class room, and one additional session on NSSI. Parents and school staff receive an online psychoeducation on NSSI. School health care personnel receive a 2-day workshop on NSSI and suicidality.
  Arms: Addressing NSSI in schools
Other: Control condition — Participating adolescents, parents, teachers and health care personnel receive no intervention during four months
  Arms: Control condition

SUMMARY:
The aim of this study is to study the effectiveness of a whole-school approach that addresses non-suicidal self-injury and targets adolescents, parents and teachers. Whether training and interventions can influence NSSI will be examined. Furthermore, investigations will be conducted to examine whether this whole-school approach can reduce symptoms of mental health problems in adolescents, reduce stigma och increase help-seeking and perception of social support. Using a clustered waitlist control design, six lower secondary schools were randomized to either intervention or waitlist during four months (control groups were then given the intervention). Measures of NSSI, suicidality, mental well-being, stigma, attitudes, help-seeking and perceived social support were administered at baseline, after the intervention and at 6, 12 and 18-months follow-up. Two hundred and sixty-seven adolescents in seventh and eight grade participated in the study (135 active group and 132 control group). The interventions were delivered during four months. For adolescents, interventions were delivered in the class room and consisted of five sessions of the Youth Aware of Mental Health (YAM) program and one additional session focusing specifically on knowledge, stigma and attitudes toward NSSI (KRAS). Parents were offered an online psychoeducation on NSSI, as were all school staff during this time period. School health care personnel, nurses, psychologist and counsellors and other school staff, such as teachers' aids, support staff and mentors took part in a 2-day workshop on NSSI and suicidality.

ELIGIBILITY:
Inclusion Criteria:

* being a student in grade 7 and 8 in lower secondary school

Exclusion Criteria:

* special classes for refugees recently arrived in Sweden with insufficient knowledge of the Swedish language
* special classes for adolescents with intellectual disability

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 267 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-12 (Actual)

PRIMARY OUTCOMES:
Life-time prevalence of nonsuicidal self-injury | Change from baseline at 4 months and at 6, 12 and 18 months
  Change in self-reported life-time prevalence of nonsuicidal self-injury is measured with a single-item (yes/no) from the Self-Injurious Thoughts and Behaviors Interview Self-Report Short-Form (SITBI-SR-SF).
Frequency of nonsuicidal self-injury | Change from baseline at 4 months and at 6, 12 and 18 months
  Change in self-reported frequency of nonsuicidal self-injury (NSSI) is measured with NSSI checklist from the Inventory of Statements About Self-injury (ISAS). Number of NSSI incidence is registered from 0 to the highest number that participants rate. High scores indicate more frequent NSSI.

SECONDARY OUTCOMES:
Health-related quality of life | Change from baseline at 4 months and at 6, 12 and 18 months
  Change in self-reported health-related quality of life (HRQOL) is measured with the 52-item version of the kid screen (KIDSCREEN 52), a self-report measure that measures the subjective HRQOL in children and adolescents between the ages of 8 and 18. KIDSCREEN 52 questionnaire consisted of 52 items assessing ten HRQOL dimensions. The KIDSCREEN-52 HRQOL questionnaire assesses the frequency of behavior/feelings or and use a 5-point Likert response scale. Scores are computed for each dimension and are transformed into T-values with a mean of 50 and a standard deviation of 10. Higher scores indicate higher HRQOL.
nonsuicidal self-injury expectancy | Change from baseline at 4 months and at 6, 12 and 18 months
  Change in self-reported nonsuicidal self-injury expectancy is measured with the Non-Suicidal Self-Injury Expectancy Questionnaire (NEQ), which is a self-report measure that measures attitudes and expectancy to own and others' NSSI. A shortened 10-item version was used with items scored on a 4-point Likert scale, ranging from 10 to 40, with higher scores indicating higher endorsement of NSSI expectancies.
Perceived Social Support | Change from baseline at 4 months and at 6, 12 and 18 months
  Change in self-reported perceived social support was measured using the Multidimensional Scale of Perceived Social Support, which is a self-report scale that measures perceived social support. It contains 12 items and is scored on a 7-point Likert scale with total scores ranging from 12 to 84, with higher scores indicating higher levels of perceived social support.
Stigma | Change from baseline at 4 months and at 6, 12 and 18 months
  Change in self-reported stigma is measures with the Mental Health Stigmatization Scale-Revised (PMHSS-R). PMHSS-R assess perceptions of stigma awareness and agreement related to mental-health in peers. The subscales include six and five items rated on a five-point Likert scale (1 = disagree completely, 5 = agree completely). An individual score is generated by adding up all items of each subscale, which ranges from 6 to 30 (awareness) and 5 to 25 (agreement). Higher scores indicate higher levels of stigma agreement and stigma awareness, that is, higher levels of mental health related stigmatizing attitudes.
Help-seeking | Change from baseline at 4 months and at 6, 12 and 18 months
  Change in self-reported help-seeking is measured with Help-Seeking Acceptability at School, Adult Help for Suicidal Youth and Reject Codes of Silence, which is a self-report measure that assesses attitudes toward seeking help from adults in three domains: "Help seeking acceptability", "Adult help for suicidal youth" and "Reject Codes of Silence". The total score includes 11 items which are scored on a 4-point Likert scale. Scores range from 4 to 16 (help-seeking acceptability); 3 to 12 (Adult help), and 3 to 12 (rejecting codes of silence). Higher scores indicate better outcome and a more positive attitude to help-seeking.
Suicidal ideation | Change from baseline at 4 months and at 6, 12 and 18 months
  Change in self-reported suicidal ideation is assessed with the Self-Injurious Thoughts and Behaviors Interview Self-Report Short-Form (SITBI-SR-SF) as single-item assessment of prevalence yes/no.

OTHER OUTCOMES:
Difficulties in emotion regulation | Change from baseline at 4 months and at 6, 12 and 18 months
  Changes in self-reported difficulties in emotion regulation is measures with the 16-item version of the Difficulties in Emotion Regulation Scale (DERS-16). Total scores range from 16 to 80 with higher scores indicating higher levels of difficulties in emotion regulation.
Self-criticism | Change from baseline at 4 months and at 6, 12 and 18 months
  Change in self-reported self-criticism is measures using the Self-Rating Scale (SRS), which is a self-report measure to assess self-criticism. It contains of 8 items which are scored on a 7-point Likert scale. The total scale ranges from 8 to 56 with higher scores indicating higher levels of self-criticism.

CONTACTS AND LOCATIONS:
Overall Officials: Maria A Zetterqvist, PhD, Principal Investigator — CSAN, BKV, Linköping university
Locations (1):
- Linköping university, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bjureberg J, Ljotsson B, Tull MT, Hedman E, Sahlin H, Lundh LG, Bjarehed J, DiLillo D, Messman-Moore T, Gumpert CH, Gratz KL. Development and Validation of a Brief Version of the Difficulties in Emotion Regulation Scale: The DERS-16. J Psychopathol Behav Assess. 2016 Jun;38(2):284-296. doi: 10.1007/s10862-015-9514-x. Epub 2015 Sep 14. PMID 27239096
- [Background] Hooley JM, Ho DT, Slater J, Lockshin A. Pain perception and nonsuicidal self-injury: a laboratory investigation. Personal Disord. 2010 Jul;1(3):170-9. doi: 10.1037/a0020106. PMID 22448633
- [Background] Klonsky ED, Glenn CR. Assessing the functions of non-suicidal self-injury: Psychometric properties of the Inventory of Statements About Self-injury (ISAS). J Psychopathol Behav Assess. 2009 Sep;31(3):215-219. doi: 10.1007/s10862-008-9107-z. Epub 2008 Oct 30. PMID 29269992
- [Background] McKeague L, Hennessy E, O'Driscoll C, Heary C. Peer Mental Health Stigmatization Scale: psychometric properties of a questionnaire for children and adolescents. Child Adolesc Ment Health. 2015 Sep;20(3):163-170. doi: 10.1111/camh.12088. Epub 2015 Feb 16. PMID 32680400
- [Background] Nearchou F, O'Driscoll C, McKeague L, Heary C, Hennessy E. Psychometric properties of the Peer Mental Health Stigmatization Scale-Revised in adolescents and young adults. Early Interv Psychiatry. 2021 Feb;15(1):201-205. doi: 10.1111/eip.12933. Epub 2020 Feb 9. PMID 32037717
- [Background] Nock MK, Holmberg EB, Photos VI, Michel BD. Self-Injurious Thoughts and Behaviors Interview: development, reliability, and validity in an adolescent sample. Psychol Assess. 2007 Sep;19(3):309-17. doi: 10.1037/1040-3590.19.3.309. PMID 17845122
- [Background] Ravens-Sieberer U, Gosch A, Rajmil L, Erhart M, Bruil J, Duer W, Auquier P, Power M, Abel T, Czemy L, Mazur J, Czimbalmos A, Tountas Y, Hagquist C, Kilroe J, Kidscreen Group E. KIDSCREEN-52 quality-of-life measure for children and adolescents. Expert Rev Pharmacoecon Outcomes Res. 2005 Jun;5(3):353-64. doi: 10.1586/14737167.5.3.353. PMID 19807604
- [Background] Wyman PA, Brown CH, Inman J, Cross W, Schmeelk-Cone K, Guo J, Pena JB. Randomized trial of a gatekeeper program for suicide prevention: 1-year impact on secondary school staff. J Consult Clin Psychol. 2008 Feb;76(1):104-15. doi: 10.1037/0022-006X.76.1.104. PMID 18229988
- [Background] Zetterqvist M, Lundh LG, Dahlstrom O, Svedin CG. Prevalence and function of non-suicidal self-injury (NSSI) in a community sample of adolescents, using suggested DSM-5 criteria for a potential NSSI disorder. J Abnorm Child Psychol. 2013 Jul;41(5):759-73. doi: 10.1007/s10802-013-9712-5. PMID 23344701
- [Background] Hasking P, Boyes M. The Non-Suicidal Self-Injury Expectancy Questionnaire: Factor structure and initial validation. Clinical Psychologist. 2018;22(2):251-261. doi:10.1111/cp.12127
- [Background] Zimet GD, Powell SS, Farley GK, Werkman S, Berkoff KA. Psychometric characteristics of the Multidimensional Scale of Perceived Social Support. J Pers Assess. 1990 Winter;55(3-4):610-7. doi: 10.1080/00223891.1990.9674095. PMID 2280326